CLINICAL TRIAL: NCT00250133
Title: Microbiologic Effect of Selective Decontamination of the Digestive Tract With Colistin, Gentamicin and Nystatin
Status: Terminated | Type: Observational
Why Stopped: Unable to obtain funding to complete study never started study
Sponsor: University of Pittsburgh (Other)
Other Study IDs: IRB#0503005
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2007-09-03 (Estimated); Status verified 2007-08

CONDITIONS: VRE Colonization
Keywords: selective decontamination of the digestive tract
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: Blood draws

SUMMARY:
Selective decontamination of the digestive tract (SDD) is a prophylactic measure aimed at reducing Gram negative flora in the gut with an aim to reduce nosocomial infections such as ventilator-associated pneumonia. A recent large randomized trial in the Netherlands showed that SDD use was associated with reduced mortality in the ICU. Theoretically, SDD may select for Gram positive organisms such as MRSA or VRE. This was not observed in the Dutch study, but the rates of MRSA and VRE are very low in hospitals in the Netherlands. Fears of selection of MRSA and VRE have limited application of SDD in the United States.

In this pilot study, 40 patients in the transplant intensive care unit (where SDD has been used intermittently for at least 10 years), will be randomized to SDD or no SDD. These patients will be known to be VRE positive at baseline. The effects of SDD on the density of VRE in the stool on day 7 compared to pre-SDD will be the primary endpoint. Secondary endpoints will be detection of MRSA and colistin resistant Pseudomonas in the stool.

DETAILED DESCRIPTION:
Study Design We will enroll 40 consecutive patients with VRE colonization who are admitted to Transplant ICU of Montefiore Hospital.

Methods:

A total of 40 patients will be randomized to SDD or no SDD by the Investigational Drugs Service of the Pharmacy. No placebo will be used for those assigned not to receive SDD. Patients will either receive standard of care or standard of care + SDD. No treatment of any kind is being withheld from the participants. Enrolled patients will be those known to be colonized with VRE (after obtaining informed consent from patients or patients' proxy). SDD will be given enterally through the nasogastric tube which will then be clamped for 1 hour. SDD will be stopped when patients are extubated. Otherwise SDD will be given for 7 days.

Day 1 is when patients are started on SDD which consists of colistin 100 mg, gentamicin 80mg, and nystatin 2 million/U in 23mL. It is given every 6 hour via a nasogastric tube with the nasogastric tube then clamped for 1 hour. Stool will be collected once a day at baseline (pre administration of SDD), and then days 4, 7 and 14 for quantitative culture of resistant pathogens in the stool. VRE, MRSA and Pseudomonas aeruginosa will be sought. An endotracheal aspirate once a day will also be collected on these days (baseline, 1, 4, 7, and 14) for qualitative culture for the presence of MRSA and Pseudomonas aeruginosa. If there are no bowel movements on the days that stool is to be collected, no samples will be obtained. In addition, if the endotracheal tube is pulled, no further endotracheal aspirates will be obtained. Samples will only be obtained if available.

In addition, for women of child bearing potential (any female who is biologically capable of becoming pregnant), a small sample (about 1 teaspoonful) of blood will be taken from a vein in the subject's arm for a pregnancy test, prior to study drug administration. Pregnant women, or women who are currently breast-feeding an infant, will not be allowed to take part in this study.

The primary microbiologic endpoint will be measurement of fecal density of VRE on day 7, in comparison to measurements on day 1. Secondary endpoints are changes in VRE fecal density from baseline to day 14, changes in MRSA fecal density from baseline to day 14, and presence of colistin resistant Pseudomonas in stool or endotracheal aspirates at day 14.

The following information will also be collected: Demographic data (address, date of birth, etc.) which includes age, sex, height, weight, and state of birth, previous reports associated with the participant's condition, laboratory results, current medication use, and any other prior medical problems/history. This information will be obtain from the medical record and/or the subject and become part of the research record.

Sample storage of the organism

The biologic samples (organism) will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. The biologic samples will be provided to Dr. Curtis Donskey, Case Western Reserve University, Cleveland, Ohio. Dr Donskey will perform colony counts on the samples in order to determine the density of organisms in the sample, using methods he described in work he published in the New England Journal of Medicine (11). All samples will be provided de-identified. Dr Paterson will perform pulsed field gel electrophoresis on the isolates to determine if isolates are genotypically identical between baseline and post-SDD. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in Dr Paterson's laboratory in Scaife Hall, Room 812, 3550 Terrace Street or in Donskey's laboratory at the Cleveland Veterans Affairs Medical Center, East Avenue, Cleveland OH.

ELIGIBILITY:
Inclusion Criteria:

* Patients in ICU who are identified as having VRE colonization by Infection Control's surveillance swabs or by the presence of VRE in clinical specimens.
* Patients must be above >18 years of age.
* Patients in whom there is an expectation of at least 4 days of mechanical ventilation.
* Presence of a nasogastric or enteral feeding tube.
* Written informed consent from patient or a proxy.

Exclusion criteria:

* Allergy to colistin, gentamicin or nystatin.
* Pregnancy.
* Intestinal transplant or multivisceral transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States